CLINICAL TRIAL: NCT07161622
Title: Effects of Low Level Laser Therapy Versus Muscle Energy Techniques Among Diabetic Patients With Frozen Shoulder
Brief Title: Comparing Low-Level Laser and Muscle Energy Techniques in Diabetic Frozen Shoulder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Aqsa Majeed, Dr. Aqsa Majeed, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zunaira
Record Dates: First submitted 2025-09-05; First posted 2025-09-08 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; Low-Level Laser Therapy; Muscle Energy Technique,; Range of Motion; Diabetes
MeSH Terms: conditions — Bursitis; Diabetes Mellitus | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low-Level Laser Therapy (LLLT) + Conventional Therapy (Experimental): Participants received LLLT with a Ga-Al-As diode laser (830 nm, 100 mW) applied to anterior capsule, posterior capsule, and subacromial area (4 J/cm² per site, 60-90 sec each), three times per week for 8 weeks. Along with LLLT, all participants received conventional therapy (moist heat, pendulum exercises, passive/active-assisted ROM, isometric strengthening, and postural correction training).
  Interventions: Other: Low-Level Laser Therapy (LLLT); Other: Muscle Energy Technique (MET)
- Muscle Energy Technique (MET) + Conventional Therapy (Experimental): Participants received MET for shoulder muscle groups (internal/external rotators, flexors, extensors). Each contraction was ~20% effort, held for 10 sec, followed by 5 sec relaxation and passive stretch to a new end range. Three to five cycles per group, ~20 minutes/session, three times per week for 8 weeks. Along with MET, all participants received the same conventional therapy as Arm A.
  Interventions: Other: Low-Level Laser Therapy (LLLT); Other: Muscle Energy Technique (MET)

INTERVENTIONS:
Other: Low-Level Laser Therapy (LLLT) — Participants received LLLT using a gallium-aluminium-arsenide (Ga-Al-As) diode laser device (BTL-5000, UK). The laser operated at a wavelength of 830 nm and a power output of 100 mW. Irradiation was applied at three sites (anterior capsule, posterior capsule, subacromial area) using a stationary-contact technique for 60-90 seconds each, delivering 4 J/cm² per site. Sessions were administered three times weekly for eight weeks.
  Conventional Therapy (for both groups):
  15 minutes of moist heat (Chattanooga Hydrocollator)
  Pendulum exercises
  Passive and active-assisted ROM exercises
  Isometric strengthening of rotator cuff and scapular stabilizers
  Postural correction training
Other: Muscle Energy Technique (MET) — Participants received MET for major shoulder muscles (internal/external rotators, flexors, extensors). Each contraction was performed at ~20% of maximum effort, sustained for 10 seconds, followed by 5 seconds relaxation, and then passive stretch to new end range. Three to five cycles per muscle group were performed. Sessions lasted ~20 minutes, three times weekly for eight weeks.
  Conventional Therapy (same as Arm A):
  15 minutes of moist heat
  Pendulum exercises
  Passive and active-assisted ROM exercises
  Isometric strengthening of rotator cuff and scapular stabilizers
  Postural correction training

SUMMARY:
The current study is to evaluate the comparative effects of low-level laser therapy and muscle energy technique on pain, range of motion, and functional results in diabetic patients with frozen shoulder. This research aims to enhance the existing data on managing diabetes-related musculoskeletal issues by assessing the comparative advantages of various therapies, therefore assisting physicians in choosing appropriate, patient-centred rehabilitation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants were male and female individuals aged 18 to 65 years with a verified diagnosis of type 2 diabetes mellitus and clinical manifestations of frozen shoulder for at least three months. The diagnosis was determined by limited glenohumeral joint mobility, characterised by a decrease of ≥20° in a minimum of three active movements: flexion <144°, abduction <120°, and external rotation <72°. Cases of both unilateral and bilateral nature were incorporated.

Exclusion Criteria:

* The exclusion criteria included a history of traumatic shoulder injury or prior surgery; neurological involvement, such as brachial plexus injury or cervical radiculopathy; rotator cuff tears or other ligamentous pathologies; tumours or malignancies affecting the shoulder; and corticosteroid injection within the preceding three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Shoulder function | Baseline, 4 weeks, and 8 weeks after intervention initiation.
  Measured using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, a validated patient-reported outcome measure assessing disability and symptoms related to upper limb musculoskeletal disorders. Higher scores indicate greater disability.